CLINICAL TRIAL: NCT01836159
Title: iPad Technology for HOME Rehabilitation in Patients After Stroke: iHOME Acute/Chronic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Sunnybrook Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 13-059C
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Fine Motor Function Deficit and Visual Neglect Post-stroke
Keywords: Stroke Rehabilitation; iPad; Fine Motor Function; Ischemic Stroke; Visual Neglect
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard/ Usual Care (Other): Patients may receive outpatient rehabilitation as required as part of usual/standard care. No experimental intervention will be given to this group.
  Interventions: Other: Standard/ Usual Care
- iPad Intervention (Experimental): Patients randomized to the iPad arm will be instructed to self-administer 20 minutes of game sessions per day for 10 days over a 2 week (14 day) period.
  Interventions: Other: iPad Intervention

INTERVENTIONS:
Other: iPad Intervention — Patients are to self-administer 20 minutes of gaming sessions, in any configuration that is preferred. Patients will be instructed to play the iPad game with the more affected arm/hand. Start and stop times of the iPad intervention will be downloaded from the iPad, which will allow calculation of the total "dose" received. Patients may receive outpatient rehabilitation as required as part of usual care.
  The 'Stroke Rehab' software for the iPad was specifically designed for patients with either fine motor weakness and/or neglect. It contains 6 stages:
  1. Popping a stationary balloon
  2. Popping a moving balloon
  3. Popping a pair of stationary balloons
  4. Popping a pair of moving balloons
  5. Stretching a balloon to pop
  6. Balloon/Text distraction test
  Arms: iPad Intervention
Other: Standard/ Usual Care — Patients may receive outpatient rehabilitation as required as part of usual care. Patients will be instructed not to play with an iPad during the 2 week intervention period (in case they have one).
  Arms: Standard/ Usual Care

SUMMARY:
A pilot randomized, two parallel group study comparing an iPad software game application versus standard care in post-stroke patients.

Study hypothesis: Tablet PC technology using the iPad is a feasible and potentially efficacious tool which has the potential to promote fine motor recovery of the upper extremity after stroke.

DETAILED DESCRIPTION:
The standard one hour of out-patient rehabilitation is insufficient in providing the repetitive intense training required for rehabilitation of fine motor recovery. There are also limited interventions are available for home use after discharge from a rehabilitation centre. Hence, there is now a need to determine the feasibility of innovative strategies for home use, to cover the gap after discharge from rehabilitation institutions.

iHOME is an original, low cost, potentially high impact intervention to fulfil this gap. If proven to be effective, the use of tablet technology has a broad range of potential outcomes and benefits. The anticipated public benefit is for stroke patients to be able to potentially employ the iPad, an accessible technological device, as an expansion of rehabilitation in an in-home setting.

iHOME is a pilot randomized controlled trial with a blinded outcome assessment. The trial is subdivided into iHOME Acute and iHOME Chronic, where patients have had a stroke less than 3 months or more than 6 months ago, respectively, at the time of randomization. Participants will be randomly allocated in a 1:1 ratio to the interventions arms (i.e. the investigational and control group).

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided written consent prior to entry into the study
* Males or females, 18 - 85 years of age
* Evidence of ischemic or hemorrhagic stroke confirmed by CT or MRI head scan
* Patient with onset of symptoms less than 3 months (for iHOME Acute) or patient more than 6 months (for iHOME Chronic) at the time of randomization
* Measurable deficit of the upper extremity ≥3 according to the Chedoke McMaster scale e.g. participants should be able to touch their chin and contralateral knee to be eligible (for iHome Acute), or measurable deficit of the upper extremity ≥4 according to the Chedoke McMaster scale e.g. participants should be able to touch their chin and contralateral knee to be eligible (for iHome Chronic)
* Functional independence prior to present stroke (mRS = 0-1)
* Patient is alert, medically stable according to the treating physician and able to follow simple verbal commands

Exclusion Criteria:

* Patient had stroke onset more than 3 months ago (for iHOME Acute) or patient had stroke onset less than 6 months ago (for iHOME Chronic)
* Inability to follow verbal commands or having global aphasia
* Severe illness with life expectancy less than 3 months
* Uncontrolled hypertension, unstable angina, or recent myocardial infarction
* History of seizures
* Participation in another clinical trial involving rehabilitation or investigational drug
* Unable to comply with the protocol
* Patient has any condition(s) that would warrant exclusion from the study
* Any medical condition that might confound the interpretation of results or put the patient at risk

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Total "dose" of intervention received as a proportion of the scheduled time | 10 days over a 2 week period
  The maximum total dose of intervention is 200min (20 min/day x 10 days). A 70% received intervention (≥140 min) from the total scheduled time will be considered successful. This will be measured by the amount of time the patient uses the application (this data is stored in the application).

SECONDARY OUTCOMES:
Efficacy in fine motor function skills | 3 business days after final study intervention session
  Efficacy will be measured by an improvement in the time to complete the nine-hole-peg test; the time to magnify and pop the balloons in the iPad software application as determined by the iPad score; the number of fine motor tasks that participants completed on the Wolf Motor Function Test; and an improvement on the Box and Block Test in the post-intervention visit. Efficacy in visual neglect will be measured by an improvement in the Star Cancellation or Line Bisection Test.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Schweizer, PhD, Study Director — Li Ka Shing, St Michael's Hospital; Chi-Ming Chow, MD, Study Director — Unity Health Toronto; Gustavo Saposnik, MD, MSc, Principal Investigator — Unity Health Toronto
Locations (3):
- Canada (3):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Rehabilitation Institute, Toronto, Ontario

REFERENCES:
- [Derived] Saposnik G, Chow CM, Gladstone D, Cheung D, Brawer E, Thorpe KE, Saldanha A, Dang A, Bayley M, Schweizer TA; iHOME Research Team for the Stroke Outcomes Research Canada Working Group. iPad technology for home rehabilitation after stroke (iHOME): a proof-of-concept randomized trial. Int J Stroke. 2014 Oct;9(7):956-62. doi: 10.1111/ijs.12328. Epub 2014 Jul 7. PMID 25042159